CLINICAL TRIAL: NCT02866708
Title: Acute and Long-term Clinical Effects of Intermittent Negative Pressure on Wound Healing in Spinal Cord and the Peripheral Circulation in Spinal Cord Injured Subjects
Brief Title: The Effects of Intermittent Negative Pressure on Wound Healing and Peripheral Circulation in Spinal Cord Injured Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Otivio AS (Industry)
Responsible Party: Principal Investigator, Jonny Hisdal, Dr. Jonny Hisdal, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/1318 REK sørøst D
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Wound Healing, Leg and Foot Ulcers, Macrocirculation, Microcirculation
MeSH Terms: conditions — Foot Ulcer

STUDY DESIGN:
Intervention Model Description: 16 week crossover pilot study comparing intermittent negative pressure (40mmHg) applied to the lower leg and foot plus standard best practice wound care comapred to standard best practice wound care alone.
Who Masked: Outcomes Assessor
Masking Description: Two experienced outcome assessors/outcome adjudicators (certified wound nurse or physician or wound trained health care specialist) will assess the wound photographs using Photographic wound assessment tool (PWAT 0-24 score). At least one of the PWAT assessors will be blinded to the study group's assignments, and will not be involved in the study otherwise (intervention or in the standard wound care).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intermittent negative pressure (INP) therapy (Experimental): At baseline, the participants will be randomized into 2 groups: 1) INP therapy or 2) control with no INP therapy.
  The 1) patients randomized to INP therapy will start with 8 weeks INP therapy two hours per day divided into timed sections (1-3 times per day or use the device as many times as practical for the individual as long as the total time is two hours). After 8 weeks of INP therapy, final measures will be performed at the Vascular lab before the participants starts their 8-week control period.
  Interventions: Device: Intermittent negative pressure device
- Control (No Intervention): The participants randomized to control will continue their usual wound care for 8 weeks without INP therapy. The control group will start INP therapy after 8 weeks. After 8-weeks without intervention, the participants allocated to the control-group will be asked to start with INP therapy for 8 weeks before a final examination. The participants in the control group will receive vascular assesment at baseline, week 8 (end of control).

INTERVENTIONS:
Device: Intermittent negative pressure device — This intervention study will be designed as a randomized cross-over study.
  Other Names: FlowOx™ , Pulsating negative pressure device, Oscillating negative pressure device
  Arms: Intermittent negative pressure (INP) therapy

SUMMARY:
This is a pilot study to evaluate the treatment effect of INP on wound healing and tissue perfusion for a larger randomized controlled trial (RCT). This randomized cross-over pilot study will look at the effects of intermittent negative pressure (INP) therapy wound healing and the peripheral macro- and microcirculation in spinal cord injured patients with chronic leg and foot ulcers (6 weeks or more at inclusion). The project is designed as a randomized clinical trial with single-subject multiple baseline design. We will perform convenience sampling of spinal cord injured patients with leg and foot ulcers, with the last recruitment by the end of december 2016.To ensure equal distribution of participants in each study arm, we will perform block randomization. A statistician will randomized patients to either intervention arm or control arm before start of the study: At baseline, each participants will be randomized into either A) 8 weeks without intervention OR B) 8 weeks with start INP therapy 2 hours per day divided into 2-3 timed sections. After the 8 weeks, participants in the the control group (A) will be re-examined, and start 8-week INP therapy. Also the intervention (INP) will be subjected to the same lower limb in each individual throughout the study period. The other leg will act as a intra-individual control.

At baseline (week 0), and during the course of the study (every 4th week), the participants' wounds will be measured by a wound nurse. Baseline (before start of INP therapy) and after intervention the following measures will be performed: Demographic data (weight, height, ABI), Segmental pulse-volume-recording, Segmental skin perfusion pressure with a laser Doppler sensor and a pressure cuff to evaluate reactive hyperemia (Sensilase, Väsamed) and health surveys (SF-36/EQ-5D-5L and customized wound questionnaire) or similar will be examined at baseline and and the end of the study period. Otivio AS has supplied the FlowOx devices and provided the necessary training to perform this project. Outcome variables assessed before and after the study period will be: wound healing (primary endpoint), quality of life (secondary endpoint), skin perfusion pressure (secondary endpoint), ankle-brachial pressure (secondary endpoint) and segmental pulse-volume recording (secondary endpoint). The aim of this project is to prospectively examine and elucidate the effect of intermittent negative pressure therapy applied to a limited part of the lower limb on clinically relevant measures related to wound healing and peripheral macro- and microcirculation in patients with spinal cord injury.

The hypotheses of the study are:

* Application of INP in patients with spinal cord injury, by the use of the FlowOx™ device, will improve wound healing in the foot compared to before treatment (baseline) and compared to standard wound care alone.
* Application of INP in patients with spinal cord injury, by the use of the FlowOx™ device, will improve macro- and microcirculation in the foot compared to before treatment (baseline) and compared to standard wound care alone in patients with spinal cord injury.
* Application of INP in patients with spinal cord injury, by the use of the FlowOx™ device, will improve macro- and microcirculation in the intervention foot compared to the control foot and compared to standard wound care alone in patients with spinal cord injury.

ELIGIBILITY:
We will perform convenience sampling of spinal cord injured patients with leg ulcers, recruited through health professionals affiliated with Sunnaas Rehabilitation hospital.

Inclusion Criteria:

* Able and willing to provide informed consent
* Age: 18-96 years
* Affected foot/shoe size <46 (approximate foot length< 29,5 cm)
* Spinal cord injury preferably with a non-healing leg/foot ulcer/pressure wound for more than 6 weeks

Exclusion Criteria:

* Incapable to consent voluntarily, i.e. patients who are not able to consent due to their mental status, or who are not willing or able to perform the negative pressure therapy in a sitting position
* Not adhering to the INP therapy program
* Patients with an expected life-span less than 3 months
* Patients in which a deep venous thrombosis or pulmonary embolism is suspected
* Bilateral amputation of lower extremity

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Percentage change in wound healing after 8 weeks of control and after 8 weeks of INP therapy | 16 weeks (baseline and after 8 and 16 weeks
  Measurement of healing to provide a means by which progress over time to wound closure can be identified. A wound nurse will take pictures at study start and at follow-up. Photographs will be measured and analysed using the ImageJ software. Reference: Schneider, C. A.; Rasband, W. S. & Eliceiri, K. W. (2012), "NIH Image to ImageJ: 25 years of image analysis", Nature methods 9(7): 671-675, PMID 22930834
Photographic wound assessment tool, PWAT 0-24 score | 16 weeks (baseline and after 8 and 16 weeks
  PWAT is wound assessing tool consisting of 6 domains that assess the composition of the wound bed and viability of the wound edge and periulcer skin that are capable of being viewed using a wound photograph. hese six domains include wound edges, necrotic tissue type and amount, skin color surrounding wound, granulation tissue type, and epithelialization. Scores assigned on a scale of 0 to 4 to each of the domains of the PWAT are summed to derive a total PWAT score between 0 and 24, with zero representing a completely healed ulcer. Reference: Houghton PE, Kincaid CB, Campbell KE, et al. Photographic assessment of the appearance of chronic pressure and leg ulcers. Ostomy/Wound Management. 2000;46(4):20-30

SECONDARY OUTCOMES:
Change in Quality of life (SF-36 ) after 8 weeks of control and after 8 weeks of INP therapy | 16 weeks (8 weeks intervention+8 weeks control)
Change in Segmental Skin Perfusion Pressure (SPP) after 8 weeks of control and after 8 weeks of INP therapy | 16 weeks (8 weeks intervention+8 weeks control)
  Multiple levels can be assessed on limbs; bilateral measurement helps to manage test time. Not susceptible to interference effects from medial calcification Requires use of pressure cuffs to occlude blood flow for specified time period in order to evaluate reactive hyperemic response to controlled release of pressure. Graphical output of pressure and perfusion during cuff deflation indicates the pressure (mmHg) at which skin perfusion is found to return in addition to pressure contour.
Change in Pulse Volume Recording (PVR) after 8 weeks of control and after 8 weeks of INP therapy | 16 weeks (8 weeks intervention+8 weeks control)
  PVR shows variations in the volume of blood passing through a limb during each cardiac cycle. The instrument that will be used to measure PVR for this study is Sensilase (Vasamed, USA) OR MacroLab (STR Teknikk, strteknikk.no, Aalesund, Norway).
  Multiple levels can be assessed on limbs. The measures are not susceptible to interference effects from medial calcification.
Change in Ankle-Brachial Pressure Index (ABPI) after 8 weeks of control and after 8 weeks of INP therapy | 16 weeks (8 weeks intervention+8 weeks control)
  The ratio of the blood pressure at the ankle (dorsal pedis artery/posterior tibial artery) to the blood pressure in the upper arm (brachial artery)
Change in Quality of life (EQ-5D-5L) ) after 8 weeks of control and after 8 weeks of INP therapy | 16 weeks (8 weeks intervention+8 weeks control)

CONTACTS AND LOCATIONS:
Overall Officials: Jonny Hisdal, PhD, Principal Investigator — Oslo University Hospital - Aker
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesodden, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Yes